CLINICAL TRIAL: NCT04134156
Title: Weight Loss and Change in Ghrelin and GLP-1 Levels After Sleeve Gastrectomy and One-anastomosis Gastric Bypass: a Randomized Clinical Trial
Brief Title: Sleeve Gastrectomy Versus One-anastomosis Gastric Bypass: Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mansoura105
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy (Active Comparator): 5-port standard sleeve gastrectomy was conducted
  Interventions: Procedure: sleeve gastrectomy
- one anastomosis gastric bypass (Active Comparator): 5-port standard one-anastomosis gastric bypass was performed
  Interventions: Procedure: one anastomosis gastric bypass

INTERVENTIONS:
Procedure: sleeve gastrectomy — 5-port sleeve gastrectomy
  Arms: Sleeve gastrectomy
Procedure: one anastomosis gastric bypass — 5-port one anastomosis gastric bypass
  Arms: one anastomosis gastric bypass

SUMMARY:
Hormonal changes after SG and OAGB involve alterations in the levels of many enteric hormones, among these hormones are ghrelin and glucagon-like peptide-1 (GLP-1). Ghrelin is an orexigenic hormone that stimulates food intake and has a documented role in the development of obesity. While ghrelin levels decrease significantly after SG as the fundus, which is the main source of that hormone, is completely removed, they tend to increase after OAGB GLP-1 plays an important role in glucose homeostasis via affecting food intake and satiety. It enhances insulin secretion, stimulates the proliferation and growth of pancreatic beta cells, inhibits food and water intake, and promotes satiety. Some studies reported that both OAGB and SG are followed by increased GLP-1 levels. We conducted this randomized study to compare SG and OAGB with regards to weight loss, comorbidity resolution, changes in ghrelin and GLP-1 hormones, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders with morbid obesity (defined as BMI > 40 kg/m2 or > 35 Kg/m2 with at least one associated comorbidity) were included. Patients who underwent previous surgery for morbid obesity were also included.

Exclusion Criteria:

* patients ageing more than 60 years
* patients with endocrine disorders
* patients with psychiatric disorders that influence perception of the study protocol
* patients unfit for general anesthesia.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
excess weight loss | 12 months after surgery
  the percentage of excess weight loss after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided